CLINICAL TRIAL: NCT04254328
Title: The Effectiveness of Nintendo Wii Fit and Inspiratory Muscle Training in Older Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cihan KILIC, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28/06/2019-908
Record Dates: First submitted 2019-12-30; First posted 2020-02-05 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure; Older People
Keywords: heart failure; older; physical activity; inspiratory muscle training; nintendo
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nintendo Wii Fit (Experimental): Nintendo Wii Fit group work program; 13 exercises in 5 groups including 3 yoga exercises, 3 balance exercises, 2 aerobic, 2 training plus exercises and 3 muscle-workout will be done respectively. Patients in this group will exercise for 8 weeks, 3 days in a week and 40-50 minutes of exercise within resting interval.
  Interventions: Device: Nintendo Wii Fit
- Respiratory (Experimental): Respiratory training group participants' will do deep breathing exercise against resistance of 30% of intraoral pressure. This exercise will be applied for 8 weeks, each day of the week, twice in a day for 15 minutes and 4-5 normal breaths after 4-5 deep breaths. Each week, intraoral pressure will be measured and new training intensity values will be determined.
  Interventions: Device: Threshold IMT
- Control (No Intervention): Patients in the control group will not be included in any exercise program, but all groups will be advised of walking in order to increase physical activity level.

INTERVENTIONS:
Device: Nintendo Wii Fit — Nintendo Wii Fit group will perform including a series of yoga, balance, aerobics and muscle workout exercises by providing visual feedback on the TV screen with the Nintendo wii fit plus game console. Patients will perform these exercises in a room allocated to the thesis supervisor and together with the thesis supervisor physiotherapist. This process takes 40-50 minutes. Before starting test and after test, weight, blood pressure, pulse, respiratory rate, oxygen saturation value will be recorded. Patients will be rested if necessary during exercise.
  Arms: Nintendo Wii Fit
Device: Threshold IMT — Patients in the breathing exercise group will perform deep breathing exercises at home by a small breathing apparatus called as Threshold IMT. It has no unexpected side effects.Patients will do this exercise twice in a day ; morning and evening during 15 minutes. After 4-5 deep breath, patients will take normal breath till feeling relaxed.
  Arms: Respiratory

SUMMARY:
Heart failure is a multisystem syndrome characterized by the body's inability to pump or increase the filling pressures required for pumping the blood needed. Typically it shows objective evidence of dyspnea and fatigue during rest or exercise, or swelling of the ankles and cardiac dysfunction. This leads to great loss of functional status and quality of life. These patients seem to be more difficult to participate in cardiac rehabilitation programs due to their more comorbid, fragile and low functional capacity. It has been shown that inspiratory muscle training, which is a part of cardiac rehabilitation, not only improves lung problems but also increases functional capacity and balance, strength of respiratory and peripheral muscles, and decreases perception of depression and dyspnea in patients. Video games are increasingly being used as an alternative to traditional rehabilitation-based exercises to improve daily activity levels and increase physical fitness in the elderly because of their recreational and motivational effects. Although Nintendo wii fit gives similar results with traditional rehabilitation practices, it causes less energy costs. This suggests that it can be a suitable rehabilitation tool for elderly people with low energy levels. A review showed that video games are safe and feasible in the elderly with heart failure. Participants' balance, cognitive functions, quality of life improved and depressive mood decreased. Video games also make older people to communicate better with other family members. The aim of this study was to investigate the effectiveness of inspiratory muscle training and nintendo wii fit exercise training in elderly patients with heart failure and to compare these practices with each other.

DETAILED DESCRIPTION:
NAME OF THE RESEARCH: The Effectiveness of Inspiratory Muscle Training and Nintendo Wii Fit Applications in Elderly Patients with Heart Failure

JUSTIFICATION AND BASIS OF THE RESEARCH: Heart failure is a multisystem syndrome characterized by the body's inability to pump or increase the filling pressures required for pumping the blood needed by the body above normal. Typically it shows objective evidence of dyspnea and fatigue during rest or exercise, or swelling of the ankles and cardiac dysfunction. This leads to great losses in the functional status and quality of life of the patients. These patients seem to be more difficult to participate in cardiac rehabilitation programs because they are more comorbid, brittle, and have low functional capacity. It has been shown that inspiratory muscle training which is a part of cardiac rehabilitation, not only improves lung problems but also increases functional capacity and balance, strength of respiratory and peripheral muscles, and decreases perception of depression and dyspnea in patients. Video games are increasingly being used as an alternative to traditional rehabilitation-based exercises to improve daily activity levels and increase physical fitness in the elderly. Although Nintendo wii fit gives similar results with traditional rehabilitation practices, it causes less energy costs. This suggests that Nintendo wii fit can be a suitable rehabilitation tool for the elderly with low energy levels. A review showed that video games are safe and feasible in the elderly with heart failure. Participants' balance, cognitive functions, quality of life improved and participants depressive mood decreased. In addition, video games enabled older people to communicate better with other family members. In the literature review, cardiac rehabilitation was found in patients with heart failure in various studies, but these applications were performed with treadmill and bicycle ergometer. There are no studies comparing the effectiveness of nintendo wii fit plus with inspiratory muscle training.

PURPOSE OF THE RESEARCH: The aim of this study is to investigate the effectiveness of inspiratory muscle training and nintendo wii fit plus exercise training in elderly patients with heart failure and to compare these practices with each other.

EXPECTED RESULTS: The first expected result of this study is that elderly patients with heart failure accept inspiratory muscle training and Nintendo wii fit plus video game as a rehabilitation tool. If patients adopt these two rehabilitation modalities as an alternative to standardized cardiac rehabilitation instruments such as bicycle ergometers and treadmills, the content and availability of home-based cardiac rehabilitation will be increased. The video game group participants will be performed in the hospital environment and under the supervision of a physiotherapist but exergame could be a home based rehabilitation application when necessary safety precautions are taken and appropriate patient selection is made. When the practices in this study are adopted by the patients, their participation in rehabilitation and physical activity will be higher and hospital visits and thus medical costs will be reduced as the content of home-based rehabilitation increases. Video games have been shown to make family members closer to each other. Thus, this study will provide not only medical and physical capacity, but also psychological and social benefits. Investigators believe that statistically significant results from this study will inspire physical, functional, emotional, emotional and social improvement studies among other elderly people who have different medical problems.

DESIGN OF THE RESEARCH: This is a prospective, experimental, before and after research. In this study, randomization will be performed first. 45 patients will be randomized into 3 columns in the microsoft excel program.

DESCRIPTION OF THE WORKING GROUP: The population of this study consisted of patients aged 60 years and older who were followed up and treated with the diagnosis of heart failure in Istanbul University-Cerrahpaşa Cardiology Institute. "Timed Up and Go Test", which is one of the tests to be performed for these patients, the number of samples was found to be 45 with 95% confidence level and 80% power.

Inclusion criteria for volunteers:

* 60 years and older
* individuals who can walk (even with the help of any device)
* individuals without visual and auditory impairment
* individuals who are cognitive to understand commands
* individuals with stable medical condition
* individuals who signed the informed consent form

Exclusion criteria for volunteers:

* Below 60 years
* individuals who cannot walk (even with the help of any device)
* individuals with visual or auditory impairment
* Myocardial infarction in the last 3 months
* previous ischemic attack
* severe cognitive impairment
* serious musculoskeletal disorders
* symptomatic medical conditions that prevent exercise (pulmonary, cardiovascular, cancer, psychiatric, etc.)

VOLUNTEER SAFETY: The study will be conducted with 3 groups of patients. The respiratory group shall perform a deep breathing exercise at home through a small breathing apparatus,Threshold IMT. Threshold IMT has no unexpected side effects. The nintendo group participants will perform a number of balance exercises with the nintendo wii fit plus game console, providing visual feedback on the TV screen. The nintendo group participants will perform these exercises in a room allocated to the thesis supervisor within Istanbul University-Cerrahpaşa Institute of Cardiology and together with the supervisor physiotherapist. Blood pressure, heart rate and oxygen saturation of the patients will be monitored at the beginning of the exercises and at other times when necessary. Participants' body weight,exergame scores,expected total kilocalorie values will be also noted. The relevant hospital staff will be informed of any negative risks that may occur during or after the exercises. The place where patients will perform assessment and balance training is a hospital environment and the necessary equipment is available. All groups will be advised of physical activity such as walking.

RESEARCH PROTOCOL: Istanbul University-Cerrahpasa, Cardiology Institute in a period of 1 year ; 45 patients, 15 of the respiratory group, 15 of the nintendo group, 15 of the control group will be randomized. All patients will initially done comprehensive geriatric evaluation. The same evaluation will be repeated at the end of the 8th week. Respiratory training group programme were described after measuring intraoral pressure with the intraoral pressure measuring device. Respiratory training group participants' will do deep breathing exercise against resistance of 30% of intraoral pressure. This exercise will be applied for 8 weeks, each day of the week, twice in a day for 15 minutes and 4-5 normal breaths after 4-5 deep breaths. Each week, intraoral pressure will be measured and new training intensity values will be determined. 13 exercises in 5 groups including 3 yoga exercises, 3 balance exercises, 2 aerobic, 2 training plus exercises and 3 muscle-workout will be done respectively.

Patients in this group will exercise for 8 weeks, 3 days in a week and 40-50 minutes of exercise within resting interval.

DATA COLLECTING: Collection of data will be done by recording under observation, answering via interviewer, questionnaire and

1. Body composition measurement with BIA (Bioelectrical Impedance Analysis) weighing device,
2. Hand grip strength measurement with Hand Dynamometer,
3. Measurement of respiratory muscle strength with electronic Intraoral Pressure Measurement Device.
4. Respiratory Function Test Device .

STATISTICAL METHODS TO BE USED: Statistical analysis of the data will be performed with the Statistical Package of Social Sciences (SPSS 21) program. Min-max control will be performed after transferring the data obtained from the research to the computer. Quantitative variables will be expressed as mean and standard deviation (± ss) and qualitative variables as percentages (%). All analyzes are within the 95% confidence interval and a value of α = 0.05 will be chosen as the level of error. Shapiro-Wilk test will be used to determine whether the data are suitable for normal distribution. Paired-t test will be used for intra-group comparisons and Student-T test will be used for comparisons between groups. For non-normal distribution values, Wilcoxon test will be used for intra-group comparisons and "Mann-Whitney U test arası will be used for intergroup comparisons. For categorical data, chi-square test (χ²) will be used for the significance test of the difference between two groups in independent groups. In the comparison according to time within the group, the normally distributed data in the 3-measure data will be vary analysis of variance in repeated measures "and the" Friedman test için for non-normally distributed data will be applied. The effect size of the intra-group changes will be calculated using the formula (difference between measurements / standard deviation of the first measurement). The effect size will be interpreted 0.20-0.50 as "small,, 0.51-0.80 as" medium, and 0.81 and above as "large".

RESEARCH TESTS:

1. Socio-demographic information
2. Anthropometric measurements
3. SPPB (Short Physical Performance Battery)
4. ADL (Activities of Daily Living)
5. IADL (Instrumental Activities of Daily Living)
6. MNA-SF (Mini Nutritional Assessment Questionnaire - Short Form)
7. FRAIL (Frailty Scale)
8. SARC-F (Sarcopenia Screening Questionnaire)
9. SNAQ (Simplified Nutrition Appetite Questionnaire)
10. GDS-SF (Geriatric Depression Scale Short Form)
11. EQ-5D Quality of Life Scale
12. GAD-7 (Generalized Anxiety Disorder Test)
13. Mini-COG (Cognitive Status Test)
14. Clock Driving Test
15. Minnesota Heart Failure and Life Survey
16. Modified Medical Research Council (mMRC) Dyspnea Scale
17. Functional Ambulation Scale (FAS)
18. 6 Minutes Walk Test

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* individual who can walk (even with the help of any device)
* an individual without visual and auditory impairment
* an individual who is cognitive to understand commands
* Stable individual with medical condition
* the individual signing the informed consent form

Exclusion Criteria:

* under 60 years
* the person who cannot walk (even with the help of any device)
* with visual or auditory impairment
* MI in the past 6 months
* previous ischemic attack
* severe cognitive impairment
* serious musculoskeletal disorders
* symptomatic medical conditions that prevent exercise (pulmonary, cardiovascular, cancer, psychiatric, etc.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
The six-minute walk test (6MWT) | 0-8 weeks
  6MWT is used to determine functional exercise capacity, assess treatment efficacy, predict prognosis. This test is applied in a certain length corridor with the start and end point during 6 minute-walk. Before the test, patient is seated in a chair and rest for 10 minutes. Resting blood pressure, pulse, oxygen saturation value, dyspnea and fatigue score is recorded before and immediate after test. Before starting to test, patient is warned to tell if any problem is seen such as dizziness, pain, cramp. The patient is then asked to walk at a fast pace with a supervisor for 6 minutes. If the patient has a significant problem such as dizziness, pain, palpitation , the test is terminated immediately. At the end of test, how many meters the patient has walked for 6 minutes has recorded.
The Timed Up and Go test (TUG) | 0-8 weeks
  The Timed Up and Go test is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time it takes for a person to get out of the chair, walk three meters, turn around, return to the chair and sit down.
The Short Physical Performance Battery Test (SPPB) | 0-8 weeks
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Prof Dr, Study Director — Istanbul University-Cerrahpasa Institute of Cardiology
Locations (1):
- Istanbul University-Cerrahpasa Institute of Cardiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If the target participant is not reached, the working order can be changed.

REFERENCES:
- [Background] Kaminsky LA, Tuttle MS. Functional assessment of heart failure patients. Heart Fail Clin. 2015 Jan;11(1):29-36. doi: 10.1016/j.hfc.2014.08.002. Epub 2014 Sep 23. PMID 25432472
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Rodriguez-Pascual C, Paredes-Galan E, Ferrero-Martinez AI, Gonzalez-Guerrero JL, Hornillos-Calvo M, Menendez-Colino R, Torres-Torres I, Vilches-Moraga A, Galan MC, Suarez-Garcia F, Olcoz-Chiva MT, Rodriguez-Artalejo F. The frailty syndrome is associated with adverse health outcomes in very old patients with stable heart failure: A prospective study in six Spanish hospitals. Int J Cardiol. 2017 Jun 1;236:296-303. doi: 10.1016/j.ijcard.2017.02.016. Epub 2017 Feb 8. PMID 28215465
- [Background] Bosnak-Guclu M, Arikan H, Savci S, Inal-Ince D, Tulumen E, Aytemir K, Tokgozoglu L. Effects of inspiratory muscle training in patients with heart failure. Respir Med. 2011 Nov;105(11):1671-81. doi: 10.1016/j.rmed.2011.05.001. Epub 2011 May 31. PMID 21621993
- [Background] Bonnechere B, Jansen B, Omelina L, Van Sint Jan S. The use of commercial video games in rehabilitation: a systematic review. Int J Rehabil Res. 2016 Dec;39(4):277-290. doi: 10.1097/MRR.0000000000000190. PMID 27508968
- [Background] Griffin M, Shawis T, Impson R, Shanks J, Taylor MJ. Comparing the Energy Expenditure of Wii Fit()-Based Therapy Versus Traditional Physiotherapy. Games Health J. 2013 Aug;2(4):229-34. doi: 10.1089/g4h.2012.0078. Epub 2013 Jul 23. PMID 26192226
- [Background] Verheijden Klompstra L, Jaarsma T, Stromberg A. Exergaming in older adults: a scoping review and implementation potential for patients with heart failure. Eur J Cardiovasc Nurs. 2014 Oct;13(5):388-98. doi: 10.1177/1474515113512203. Epub 2013 Nov 6. PMID 24198306